CLINICAL TRIAL: NCT01473290
Title: A Phase III, Randomized, Double-Blind Placebo Controlled Study of the Probiotic Preparation VSL#3® Versus Placebo in the Prevention of Acute Enteritis in Patients Receiving Concurrent Chemotherapy and Pelvic Radiation Therapy
Brief Title: Probiotic Therapy in Preventing Gastrointestinal Complications in Patients Undergoing Chemotherapy and Pelvic Radiation Therapy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not activated.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N10CB; NCI-2011-03636 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000716291 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Cognitive/Functional Effects; Constipation, Impaction, and Bowel Obstruction; Diarrhea; Fatigue; Gastrointestinal Complications; Psychosocial Effects of Cancer and Its Treatment; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: diarrhea; constipation, impaction, and bowel obstruction; gastrointestinal complications; fatigue; psychosocial effects of cancer and its treatment; cognitive/functional effects; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Constipation; Intestinal Obstruction; Diarrhea; Fatigue

ARMS (2):
- Arm I (Experimental): Patients receive live freeze-dried lactic acid bacteria probiotic (VSL#3®) orally (PO) 3 times a day during RT (5-8 weeks) and for 2 weeks after completion of RT.
  Interventions: Dietary Supplement: live freeze-dried lactic acid bacteria probiotic
- Arm II (Placebo Comparator): Patients receive placebo PO 3 times a day during RT (5-8 weeks) and for 2 weeks after completion of RT.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: live freeze-dried lactic acid bacteria probiotic — Given orally (PO)
  Arms: Arm I
Other: placebo — Given PO
  Arms: Arm II

SUMMARY:
RATIONALE: Probiotic therapy may reduce or prevent gastrointestinal complications in patients undergoing chemotherapy and pelvic radiation therapy.

PURPOSE: This randomized phase III trial is studying how well probiotic therapy works in preventing gastrointestinal complications in patients undergoing chemotherapy and pelvic radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether live freeze-dried lactic acid bacteria probiotic (VSL#3®) is effective in reducing the acute treatment-related bowel function disturbances, as measured by the FACIT-D diarrhea subscale score in patients receiving concurrent chemotherapy and pelvic RT as adjuvant or primary treatment for malignancy.

Secondary

* To determine whether VSL#3® can reduce chronic treatment-related bowel dysfunction following completion of therapy.
* To examine whether VSL#3® appears to have an impact on disease-free survival.
* To bank blood products for future studies. (exploratory)
* To characterize changes in the fecal microbiota and examine for correlation with treatment assignment and symptom scores. (exploratory)

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to site of primary tumor (rectum/anus vs other), history of anterior resection of the rectum (yes vs no), total planned cumulative dose (including boost of external-beam radiotherapy [RT] or brachytherapy) (4,500-5,350 cGy vs > 5,350 cGy), and use of intensity-modulated RT [IMRT] for pelvic RT (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive live freeze-dried lactic acid bacteria probiotic (VSL#3®) orally (PO) 3 times a day during RT (5-8 weeks) and for 2 weeks after completion of RT.
* Arm II: Patients receive placebo PO 3 times a day during RT (5-8 weeks) and for 2 weeks after completion of RT.

Patients self-report symptoms using the FACIT-D, PBFQ, PRO-CTCAE, and Uniscale/fatigue weekly during RT, for 2 weeks after completion of RT, and at 12 months following the completion of RT.

Blood and stool samples may be collected from some patients for correlative studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current diagnosis of cancer that supports the use of continuous definitive or adjuvant external-beam radiotherapy (RT) to the pelvis to a minimum dose of 4,500 cGy with the following parameters:

  * The pelvis must be encompassed by the planned RT fields

    * The superior border may not lie inferior to the most inferior aspect of the sacroiliac joints
    * Portions of the rectum may have special blocking, depending upon disease site
  * The total prescription dose must lie between 4,500-5,350 cGy (inclusive)

    * A boost to primary tumor or tumor bed may be planned
  * Planned treatment is to be given 4-5 times per week on a one- treatment-per-day basis

    * The daily prescribed dose must lie between 170-210 cGy (inclusive) per day
  * No planned split-course RT
  * No proton RT
* Will receive concurrent administration of chemotherapy (fluorouracil, capecitabine, cisplatin, oxaliplatin, carboplatin, and/or mitomycin C) during pelvic RT
* No current or prior metastases beyond regional lymph nodes

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) of 0, 1, or 2
* Life expectancy ≥ 6 months
* Able to complete questionnaire(s) by themselves or with assistance
* Not pregnant or nursing
* Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only
* Fertile patients must use effective contraception
* Hemoglobin > 10.0 g/dL
* White blood cells (WBC) > 3,500/mm³
* Absolute neutrophil count (ANC) > 1,500/mm³
* Platelet count > 100,000/mm³
* Willing to abstain from ingestion of yogurt products and/or any product containing probiotics during study drug treatment
* No known allergy to a probiotic preparation
* No history of inflammatory bowel disease
* No ≥ grade 3 diarrhea, ≥ grade 3 rectal bleeding, abdominal cramping, or incontinence of stool ≤ 7 days prior to registration
* No medical condition that may interfere with ability to receive protocol treatment
* No history of gastrointestinal or genitourinary obstruction or porphyria
* No history of irritable bowel syndrome (IBS)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior abdominal-perineal resection, Hartmann procedure, or other surgical procedure leaving the patient without a functioning rectum
* No planned use of leucovorin
* No prior pelvic RT
* No use of probiotics ≤ 2 weeks prior to registration
* No use of antibiotics ≤ 3 days prior to registration
* No planned continuous antibiotic treatment during RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Average area under the curve (AUC) of the FACIT-D diarrhea subscale score assessed weekly during treatment and for two weeks following the completion of RT | Up to 12 months

SECONDARY OUTCOMES:
Bowel function measures as assessed by the clinician using the CTCAE version 4 and as assessed by the PBFQ and the PRO-CTCAE | Up to 12 months
Psychometric evaluation of the reliability and validity of the FACIT-D diarrhea subscale, PBFQ, and PRO-CTCAE | Up to 12 months
Disease-free survival | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Miller, MD, Principal Investigator — Mayo Clinic